CLINICAL TRIAL: NCT04960098
Title: Patient-Reported Outcome Measures in Patient Underwent Total Hip and Knee Arthroplasty in Galeazzi Orthopaedic Institute Milano
Brief Title: Patient-reported Outcome Measures in Patient Underwent Total Hip and Knee Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: PROMS
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis; Prosthesis Survival
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Prosthesis Failure | interventions — Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient underwent hip and knee arthroplasty: Patients with hip and knee osteoarthritis underwent hip and knee arthroplasty included in inclusion criteria.
  Interventions: Procedure: arthroplasty

INTERVENTIONS:
Procedure: arthroplasty — patient with hip and knee osteoarthritis underwent hip and knee arthroplasty

SUMMARY:
Registry of Galeazzi Orthopedic Institute: provides for the regular and systematic collection of all data (clinical and some PROMs) obtained from patients undergoing hip and knee arthroplasty to which questionnaires are proposed investigating the specific functional sphere of the joints undergoing surgery (Knee injuryOsteoarthritisOutcomeScore (KOOS-PS) and Hip injuryOsteoarthritisOutcomeScore (HOOS-PS) but also the sphere of general health (ShortForm health survey-12 (SF-12) and VisualAnalogueScale (VAS)) , in addition, of course, to the satisfaction rate.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age more than 18
* patient underwent hip or knee arthroplasty

Exclusion Criteria:

* age less than 18
* comorbidity that can results in the difficulty to come back for the follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients underwent hip and knee arthroplasty included in inclusion criteria
Sampling Method: Probability Sample
Enrollment: 5816 (Estimated)
Dates: Start 2016-01-12 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
outcome measurements | pre operative to 10 years
  improve evaluation of hip and knee arthroplasty monitoring patient reported outcome measurements before and after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided